CLINICAL TRIAL: NCT00920608
Title: A Phase I, Multi-centre, Open-label, Fixed-sequence Study to Assess the Pharmacokinetics of Methotrexate Alone and When Co-administered With AZD9056 in Subjects With Rheumatoid Arthritis
Brief Title: A Study to Assess the Pharmacokinetics of Methotrexate Given With and Without AZD9056 in Rheumatoid Arthritis Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D1520C00027
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Rheumatoid Arthritis
Keywords: AZD9056; Pharmacokinetics; interaction; Methotrexate; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — AZD9056; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): AZD9056 400 mg and Methotrexate
  Interventions: Drug: AZD9056; Drug: Methotrexate

INTERVENTIONS:
Drug: AZD9056 — Tablets for oral use. 400 mg once daily for 7 days
Drug: Methotrexate — Tablet for oral use.7.5 to 20 mg single dose administration at visit 2 and 3.
  Other Names: Various brands used

SUMMARY:
The main aim of this clinical study is to investigate whether the blood concentration of methotrexate changes when AZD9056 is co- administered together with methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with rheumatoid arthritis
* Currently on Methotrexate treatment
* Provision of informed consent

Exclusion Criteria:

* History of malignancy (except for treated squamous and basal cell carcinoma of the skin more than 5 years prior to entry)
* Patients who were taking prescription of medications listed below:

Medications that are hepatic enzyme inducers and that were inhibitors of cytochrome P450, Lovastatin

* Leflunomide, hydroxychloroquine, cyclosporin or anti-tumour necrosis factor therapies within 90 days of Visit 1, or treatment with rituximab within 1 year before Visit 1

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-05; Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of AZD9056 and Methotrexate | Pharmacokinetic samples for Methotrexate taken at baseline and and at steady state.Pharmacokinetc samples for AZD9056 taken at steady state

SECONDARY OUTCOMES:
Pharmacokinetics of AZD9056 and 7-OH Methotrexate | Pharmacokinetics samples for 7-OH Methotrexate taken at baseline and and at steady state.Pharmacokinetc samples for AZD9056 taken at steady state
Safety and tolerability (Physical examination, vital signs, electrocardiogram (ECG), safety laboratory,adverse events.) | During the whole study